CLINICAL TRIAL: NCT05611346
Title: HYPNOsis in the Management of Atopic Dermatitis in Children and Teenagers : Study Protocol of a Pilot Randomized and Controlled Trial
Brief Title: HYPNOsis in the Management of Atopic Dermatitis in Children and Teenagers
Acronym: HypnoDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/CHU/15
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic education program (No Intervention)
- Therapeutic education program and Hypnosis (Experimental)
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — The experimental group will receive 2 standardized hypnosis sessions via the "superhero costume" technique performed during this collective therapeutic education program, completed by a reinforcement through the practice of self-hypnosis at home guided by the listening of an audio recording
  Arms: Therapeutic education program and Hypnosis

SUMMARY:
Atopic dermatitis (AD) is a chronic inflammatory dermatosis, common in children. It causes pruritus and skin lesions that can have a significant impact on patients' quality of life. AD can be difficult to treat because of its chronicity, demanding local care, corticophobia and the financial cost of non-reimbursed products. Patients are often looking for therapeutic alternatives. Medical hypnosis is a therapeutic alternative via hypnoanalgesia induced by direct suggestions of comfort and skin soothing and via anxiolysis, by working on stress management and self-esteem reinforcement. Four studies are interested in its action in AD and seem to show a reduction in pruritus, skin pain, an improvement in the intensity of atopic dermatitis, sleep, mood and for some a cure of AD. These results are encouraging but limited by the absence of a control group or by the small population included. Therefore, we propose in a first step to evaluate the feasibility of an hypnosis program through a pilot study, designed in the miniature format of a future, larger scale, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 17 years
* Understanding french
* Have a clinical diagnosis of mild-to-severe AD with a SCORing Atopic Dermatitis (SCORAD)
* Referred by their referring physician in the Reunionese therapeutic education program for AD provided within the atopy school of the Reunion University Hospital. - Oral consent of the child and of one of the legal representatives collected.

Exclusion Criteria:

* Children refusing to participate in the hypnosis session
* Not having the possibility to listen to an audio file,
* Already practicing self-hypnosis for their AD before inclusion,
* Having a contraindication to hypnosis (psychiatric disorders, psychosis)
* Treated by a systemic treatment for their AD.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Asses the patient recruitment rate | 24 months
  The recruitment rate is the proportion of patients recruited into the pilot study: number of patients included/number of patients to whom the study was proposed.

SECONDARY OUTCOMES:
Assess patient compliance with self-hypnosis practice | At 1 month, 3 months, and 6 months after inclusion
  Assess patients' adherence to self-hypnosis practice at home, on a self-reported basis, using an adherence log in the experimental arm by:
  * The adherence rate at M1
  * The variation in the adherence rate over time
Patient lost sight of | At 1 month, 3 months, and 6 months after inclusion
  Evaluate the rate of patient who has been lost sight of(M1, M3, M6) in both arms, measured by the proportion of patients lost sight of/number of patients included at baseline
Patient satisfaction | At 1 month, 3 months, and 6 months after inclusion
  Assess patient satisfaction with the hypnosis program in the experimental arm using a satisfaction questionnaire
Improvements to the hypnosis program | At 6 months after inclusion
  Describe possible improvements to the hypnosis program in the experimental arm at M6 through focus group interviews with a group of volunteers aged 8-11 and a group of volunteers aged 12-17.
Effectiveness | At 1 month, 3 months, and 6 months after inclusion
  Evaluate the effectiveness of a hypnosis program (exploratory)
  * On the control of atopic dermatitis ( The change in the mean AD control score, measured by the ADCT)
  * On the severity of atopic dermatitis (The change in the mean AD severity score, measured by the PO-SCORAD)
Parents' overall impression | At 1 month, 3 months, and 6 months after enrollment
  Assess parents' overall impression of their child's AD progress with the hypnosis program, via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Juliette MIQUEL, MD, Principal Investigator — CHU de la Réunion
Locations (1):
- CHU de la Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No